CLINICAL TRIAL: NCT02007434
Title: A Single Center, Double-blind, Parallel-group, Two Factor Patient-Experience Management Study of ATX-101 (Deoxycholic Acid Injection) for the Reduction of Localized Subcutaneous Fat in the Submental Area
Brief Title: Patient Experience Study of Deoxycholic Acid Injection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-13-36
Record Dates: First submitted 2013-10-30; First posted 2013-12-10 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Moderate or Severe Submental Fullness
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Deoxycholic Acid; Lidocaine; Epinephrine; Loratadine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Paradigm 1 / Deoxycholic Acid Injection (Experimental): Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, either 6 or 8 mL (based on Baseline CR-SMFRS grade 2 or 3, respectively) on Day 0 and a cold compress applied to the treatment area.
  Interventions: Drug: Deoxycholic Acid Injection; Other: Cold Compress
- Paradigm 1/ Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL injections, either 6 or 8 mL on Day 0 and a cold compress applied to the treatment area.
  Interventions: Drug: Placebo; Other: Cold Compress
- Paradigm 2 / Deoxycholic Acid Injection (Experimental): Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, either 6 or 8 mL on Day 0, topical and injectable anesthetics (lidocaine/epinephrine) and a cold compress applied to the treatment area.
  Interventions: Drug: Deoxycholic Acid Injection; Other: Cold Compress; Drug: Lidocaine / Epinephrine
- Paradigm 2 / Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL injections, either 6 or 8 mL on Day 0, topical and injectable anesthetics and a cold compress applied to the treatment area.
  Interventions: Drug: Placebo; Other: Cold Compress; Drug: Lidocaine / Epinephrine
- Paradigm 3 / Deoxycholic Acid Injection (Experimental): Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, either 6 or 8 mL on Day 0, oral antihistamine and anti-inflammatory agents (loratadine and ibuprofen), topical and injectable anesthetics and a cold compress applied to the treatment area.
  Interventions: Drug: Deoxycholic Acid Injection; Other: Cold Compress; Drug: Lidocaine / Epinephrine; Drug: Loratadine; Drug: Ibuprofen
- Paradigm 3 / Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL injections, either 6 or 8 mL on Day 0, oral antihistamine and anti-inflammatory agents, topical and injectable anesthetics and a cold compress applied to the treatment area.
  Interventions: Drug: Placebo; Other: Cold Compress; Drug: Lidocaine / Epinephrine; Drug: Loratadine; Drug: Ibuprofen
- Paradigm 4 / Deoxycholic Acid Injection (Experimental): Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, either 6 or 8 mL on Day 0, a compression chin strap, oral antihistamine and anti-inflammatory agents, topical and injectable anesthetics and a cold compress applied to the treatment area.
  Interventions: Drug: Deoxycholic Acid Injection; Other: Cold Compress; Drug: Lidocaine / Epinephrine; Drug: Loratadine; Drug: Ibuprofen; Other: Compression Chin Strap
- Paradigm 4 / Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL injections, either 6 or 8 mL on Day 0, a compression chin strap, oral antihistamine and anti-inflammatory agents, topical and injectable anesthetics and a cold compress applied to the treatment area.
  Interventions: Drug: Placebo; Other: Cold Compress; Drug: Lidocaine / Epinephrine; Drug: Loratadine; Drug: Ibuprofen; Other: Compression Chin Strap

INTERVENTIONS:
Drug: Deoxycholic Acid Injection — Formulated as an injectable solution containing deoxycholic acid at a concentration of 10 mg/mL.
  Other Names: ATX-101; Kybella
  Arms: Paradigm 1 / Deoxycholic Acid Injection; Paradigm 2 / Deoxycholic Acid Injection; Paradigm 3 / Deoxycholic Acid Injection; Paradigm 4 / Deoxycholic Acid Injection
Drug: Placebo — Phosphate buffered saline placebo for injection
  Arms: Paradigm 1/ Placebo; Paradigm 2 / Placebo; Paradigm 3 / Placebo; Paradigm 4 / Placebo
Other: Cold Compress — A cold compress was applied to the injection area for 10 minutes before dosing and for 15 minutes after dosing.
Drug: Lidocaine / Epinephrine — Lidocaine 4% topical cream applied 45 minutes prior to dosing across the area to be treated, followed by 0.4 mL SC injections of lidocaine HCl 1% / epinephrine 1:100,000 around the perimeter of the treatment area and across the treatment area in a regular pattern 25 minutes before dosing.
  Arms: Paradigm 2 / Deoxycholic Acid Injection; Paradigm 2 / Placebo; Paradigm 3 / Deoxycholic Acid Injection; Paradigm 3 / Placebo; Paradigm 4 / Deoxycholic Acid Injection; Paradigm 4 / Placebo
Drug: Loratadine — Loratadine 10 mg orally from Day -7 until Day 7
  Arms: Paradigm 3 / Deoxycholic Acid Injection; Paradigm 3 / Placebo; Paradigm 4 / Deoxycholic Acid Injection; Paradigm 4 / Placebo
Drug: Ibuprofen — Ibuprofen 600 mg at least 1 hour prior to dosing and 600 mg 3 times a day for at least 3 days after dosing.
  Arms: Paradigm 3 / Deoxycholic Acid Injection; Paradigm 3 / Placebo; Paradigm 4 / Deoxycholic Acid Injection; Paradigm 4 / Placebo
Other: Compression Chin Strap — A compression chin strap was applied 15 minutes after dosing for at least 24 hours.
  Arms: Paradigm 4 / Deoxycholic Acid Injection; Paradigm 4 / Placebo

SUMMARY:
The objectives of this study are to determine the safety of deoxycholic acid subcutaneous (SC) injections in the submental area and to evaluate the effects of four interventions, relative to placebo in the submental area, particularly with regard to assessment and management of pain, bruising, and swelling/edema.

DETAILED DESCRIPTION:
This study evaluated the effects of four interventions, pre- and post-subcutaneous injections of deoxycholic acid injection relative to placebo in adults with submental fullness. Participants were randomized to either deoxycholic acid injection or placebo in a ratio of 4:1 and to one of four patient experience management paradigms.

Participants were required to visit the research facility on 10 separate occasions for protocol-defined treatments, procedures, tests, and observations.

ELIGIBILITY:
Inclusion Criteria:

1. Submental fat graded by the Investigator as 2 (moderate) or 3 (severe) using the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and graded by the subject as 2 (moderate amount) or 3 (large amount) using the Patient-Reported Submental Fat Rating Scale (PR-SMFRS)
2. Dissatisfaction with the appearance of the submental area expressed by the subject as a rating of 0, 1, or 2 using the Subject Self Rating Scale (SSRS)
3. History of stable body weight for at least 6 months and body mass index (BMI) of ≤ 40 kg/m².
4. Acceptable skin laxity as determined by the investigator
5. Agreement by the subject to refrain from making significant changes, in the documented judgment of the investigator, to his or her dietary or exercise habits during the course of the subject's participation.
6. Agreement to forego any treatment or behavior (e.g., unshaven facial hair)
7. Signed informed consent obtained before any study-specific procedure is performed.

Exclusion Criteria:

1. No prior intervention for submental fullness or recent cosmetic procedure in the neck or chin area
2. Absence of clinically significant health problems
3. Body mass index > 40.0 kg/m² as determined prior to randomization.
4. History of drug or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, III, MD, PhD, Study Director — Sponsor GmbH
Locations (1):
- Investigational Site, Tempe, Arizona, United States

REFERENCES:
- [Derived] Dover JS, Kenkel JM, Carruthers A, Lizzul PF, Gross TM, Subramanian M, Beddingfield FC 3rd. Management of Patient Experience With ATX-101 (Deoxycholic Acid Injection) for Reduction of Submental Fat. Dermatol Surg. 2016 Nov;42 Suppl 1:S288-S299. doi: 10.1097/DSS.0000000000000908. PMID 27787269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at one investigational center in the United States (US).
Groups:
- Paradigm 1 / Deoxycholic Acid Injection: Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, either 6 or 8 mL (based on Baseline Clinician-Reported Submental Fat Rating Scale [CR-SMFRS] grade 2 or 3, respectively) on Day 0 and a cold compress applied to the treatment area.
- Paradigm 1 / Placebo: Participants received placebo administered in 0.2 mL injections, either 6 or 8 mL on Day 0 and a cold compress applied to the treatment area.
Period: Overall Study
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Started | 17 | 4 | 17 | 4 | 16 | 4 | 18 | 4
Received Treatment | 17 | 3 | 17 | 4 | 16 | 4 | 18 | 4
Completed | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
Not Completed | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- Paradigm 1 / Deoxycholic Acid Injection: Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, either 6 or 8 mL on Day 0 and a cold compress applied to the treatment area.
- Total: Total of all reporting groups
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo | Total
Number analyzed (Participants) | 17 | 3 | 17 | 4 | 16 | 4 | 18 | 4 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.08) | 36.3 (14.05) | 42.4 (13.08) | 43.8 (11.67) | 41.3 (11.48) | 44.8 (14.84) | 42.3 (13.08) | 48.0 (8.64) | 43.5 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 1 | 11 | 2 | 10 | 3 | 9 | 3 | 51
  Male | 5 | 2 | 6 | 2 | 6 | 1 | 9 | 1 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  White | 15 | 1 | 13 | 4 | 12 | 3 | 14 | 4 | 66
  Black or African American | 1 | 2 | 3 | 0 | 2 | 1 | 3 | 0 | 12
  American Indian/Alaskan Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Weight [Mean (Standard Deviation); unit: pounds] | 191.01 (40.086) | 221.00 (34.492) | 205.61 (38.716) | 223.90 (27.534) | 205.74 (32.847) | 217.90 (11.485) | 200.30 (36.592) | 185.05 (68.356) | 202.53 (37.514)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 30.959 (4.2723) | 28.867 (4.9923) | 33.206 (4.9806) | 33.350 (3.1586) | 32.763 (3.7764) | 36.850 (2.3587) | 31.706 (3.3457) | 31.250 (7.7229) | 32.266 (4.3474)
Fitzpatrick Skin Type [Number; unit: participants] — Fitzpatrick Skin Type is a numerical classification schema for human skin color and typical response to ultraviolet (UV) light:
  * Type I: Pale white skin, blue/hazel eyes, blond/red hair; Always burns, does not tan.
  * Type II: Fair skin, blue eyes; Burns easily, tans poorly.
  * Type III: Darker white skin; Tans after initial burn.
  * Type IV: Light brown skin; Burns minimally, tans easily.
  * Type V: Brown skin; Rarely burns, tans darkly easily.
  * Type VI: Dark brown or black skin; Never burns, always tans darkly.
  participants
    I-III | 12 | 0 | 7 | 2 | 6 | 2 | 6 | 1 | 36
    IV-VI | 5 | 3 | 10 | 2 | 10 | 2 | 12 | 3 | 47
Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) [Number; unit: participants] — The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
  participants
    2 | 13 | 1 | 12 | 2 | 9 | 4 | 15 | 2 | 58
    3 | 4 | 2 | 5 | 2 | 7 | 0 | 3 | 2 | 25
Patient-Reported Submental Fat Rating Scale (PR-SMFRS) [Number; unit: participants] — The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" answered on a 5-point ordinal scale (0-4) with 0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat.
  participants
    2 | 10 | 2 | 14 | 1 | 12 | 1 | 13 | 3 | 56
    3 | 7 | 1 | 3 | 3 | 4 | 3 | 5 | 1 | 27
Subject Self Rating Scale (SSRS) [Number; unit: participants] — The SSRS assesses participant's satisfaction with their appearance in association with the face and chin on a 7-point scale from 0 to 6: where 0 = Extremely dissatisfied, 1 = Dissatisfied, 2 = Slightly dissatisfied, 3 = Neither satisfied nor dissatisfied, 4 = Slightly satisfied, 5 = Satisfied and 6 = Extremely satisfied.
  participants
    0 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 7
    1 | 8 | 1 | 9 | 3 | 10 | 3 | 8 | 1 | 43
    2 | 8 | 1 | 5 | 1 | 5 | 1 | 10 | 2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Visual Analog Scale Scores
Description: Participants were provided with a scale 100 mm in length and were asked to mark the place on the line that best represents his or her pain associated with the area treated with study drug. The scale ranged from 0 (no pain) to 100 (most severe pain possible).
Time Frame: Baseline and Day 84
Population: Safety analysis set with available data at both time points
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale | 0.0 [-2 to 5] | 0.0 [0 to 0] | 0.0 [-2 to 1] | 0.0 [0 to 0] | 0.0 [0 to 2] | 0.0 [-1 to 0] | 0.0 [-1 to 1] | 0.0 [-1 to 0]
Statistical Analysis 1: Comparison: Paradigm 1 / Deoxycholic Acid Injection vs Paradigm 2 / Deoxycholic Acid Injection; Pairwise differences between paradigms for the placebo-adjusted differences were conducted using a two-way analysis of covariance (ANCOVA) with factors for treatment, paradigm, treatment-by-paradigm interaction, and covariate of baseline CR-SMFRS score; Test type: Superiority or Other; p = 0.6803, ANCOVA; LS Mean Placebo-adjusted Difference = 0.24, 95% CI 2-sided [-0.93 to 1.41], Standard Error of Mean 0.59 — Paradigm 1 - Paradigm 2
Statistical Analysis 2: Comparison: Paradigm 1 / Deoxycholic Acid Injection vs Paradigm 3 / Deoxycholic Acid Injection; Day 0, 1 Minute. Pairwise differences between paradigms for the placebo-adjusted differences were conducted using a two-way analysis of covariance (ANCOVA) with factors for treatment, paradigm, treatment-by-paradigm interaction, and covariate of baseline CR-SMFRS score; Test type: Superiority or Other; p = 0.5206, ANCOVA; LS Mean Placebo-adjusted Difference = 0.39, 95% CI 2-sided [-0.82 to 1.60], Standard Error of Mean 0.61 — Paradigm 1 - Paradigm 3
Statistical Analysis 3: Comparison: Paradigm 1 / Deoxycholic Acid Injection vs Paradigm 4 / Deoxycholic Acid Injection; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6060, ANCOVA; LS Mean Placebo-adjusted Difference = 0.30, 395% CI 2-sided [-0.86 to 1.46], Standard Error of Mean 0.58 — Paradigm 1 - Paradigm 4
Statistical Analysis 4: Comparison: Paradigm 2 / Deoxycholic Acid Injection vs Paradigm 3 / Deoxycholic Acid Injection; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7935, ANCOVA; LS Mean Placebo-adjusted Difference = 0.15, 95% CI 2-sided [-0.98 to 1.27], Standard Error of Mean 0.56 — Paradigm 2 - Paradigm 3
Statistical Analysis 5: Comparison: Paradigm 2 / Deoxycholic Acid Injection vs Paradigm 4 / Deoxycholic Acid Injection; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9140, ANCOVA; LS Mean Placebo-adjusted Difference = 0.06, 95% CI 2-sided [-1.03 to 1.15], Standard Error of Mean 0.55 — Paradigm 2 - Paradigm 4
Statistical Analysis 6: Comparison: Paradigm 3 / Deoxycholic Acid Injection vs Paradigm 4 / Deoxycholic Acid Injection; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8754, ANCOVA; LS Mean Placebo-adjusted Difference = -0.09, 95% CI 2-sided [-1.21 to 1.04], Standard Error of Mean 0.56 — Paradigm 3 - Paradigm 4

2. Primary Outcome: Change From Baseline in Pain Assessment Using McGill Pain Questionnaire
Description: Participants rated 15 pain characteristics by using a number to signify how much of that specific type of pain they were experiencing using the Short-Form McGill Pain Questionnaire. The pain characteristic options included Throbbing, Shooting, Stabbing, Sharp, Cramping, Gnawing, Hot-burning, Aching, Heavy, Tender, Splitting, Tiring-exhausting, Sickening, Fearful, and Punishing- cruel. Participants assessed the intensity of each characteristic using the following score system: none (0), mild (1), moderate (2), and severe (3). In addition, present pain was assessed on a scale from 0 (no pain) to 5 (excruciating).
Time Frame: Baseline (predose) and Day 84
Population: Safety analysis set with available data at both time points
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Paradigm 4 / Deoxycholic Acid Injection: Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, either 6 to 8 mL on Day 0, a compression chin strap, oral antihistamine and anti-inflammatory agents, topical and injectable anesthetics and a cold compress applied to the treatment area.
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale
  Throbbing | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Shooting | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Stabbing | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Sharp | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Cramping | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Gnawing | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Hot-Burning | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Aching | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.1 (0.25) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Heavy | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.1 (0.25) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Tender | 0.0 (0.00) | 0.0 (0.00) | 0.1 (0.25) | 0.0 (0.00) | 0.1 (0.25) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Splitting | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Tiring-Exhausting | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Sickening | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Fearful | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Punishing-Cruel | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Present pain | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

3. Primary Outcome: Swelling Grading Scale Scores
Description: The following grading system was used for the assessment of swelling:
  * Swelling/edema absent (0)
  * Minimal swelling/edema contained within treatment area (1)
  * Modest swelling/edema contained within treatment area (2)
  * Substantial swelling/edema contained within treatment area (3)
  * Swelling/edema of the neck and face beyond the treatment area (4)
Time Frame: Day 84
Population: Safety analysis set with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

4. Primary Outcome: Bruising Grading Scale Scores
Description: The following grading system was used for the assessment of bruising:
  * Bruising absent (0)
  * Bruising associated with 1 to 3 needle insertion points (1)
  * Bruising spreading beyond 4 or more individual needle insertion points but contained within the treatment area (2)
  * Bruising covering the entire treatment area but contained within the treatment area (3)
  * Bruising of the neck and face beyond the treatment area (4)
Time Frame: Day 84
Population: Safety analysis set with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

5. Primary Outcome: Induration Grading Scale Scores
Description: The following grading system was used for the assessment of induration:
  * Induration absent to minimal (0)
  * Induration associated with at least approximately 30% of the treatment area (1)
  * Induration associated with greater than approximately 30% to at least 60% of the treatment area (2)
  * Induration covering the entire treatment area but contained within the treatment area (3)
  * Induration of the neck and face beyond the treatment area (4)
Time Frame: Day 84
Population: Safety analysis set with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale | 0.0 (0.00) | 0.0 (0.00) | 0.1 (0.25) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.1 (0.32) | 0.0 (0.00)

6. Secondary Outcome: Change From Baseline in Clinician-Reported Submental Fat Rating Scale (CR-SMFRS)
Description: The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Day 84
Population: Safety analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale | -0.6 (0.50) | -0.7 (0.58) | -0.6 (0.63) | -0.8 (0.96) | -0.4 (0.50) | 0.0 (0.82) | -0.4 (0.50) | -0.3 (0.50)

7. Secondary Outcome: Change From Baseline in Patient-Reported Submental Fat Rating Scale (PR-SMFRS)
Description: The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" answered on a 5-point ordinal scale (0-4) with 0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Day 84
Population: Safety analysis set with available data at both time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale | -1.2 (0.75) | -0.7 (1.15) | -0.9 (0.72) | -0.5 (1.29) | -0.8 (0.86) | -0.8 (0.50) | -0.7 (0.57) | -0.5 (0.58)

8. Secondary Outcome: Change From Baseline in Subject Self Rating Scale (SSRS)
Description: The SSRS assesses participant's satisfaction with their appearance in association with the face and chin on a 7-point scale from 0 to 6: where 0 = Extremely dissatisfied, 1 = Dissatisfied, 2 = Slightly dissatisfied, 3 = Neither satisfied nor dissatisfied, 4 = Slightly satisfied, 5 = Satisfied and 6 = Extremely satisfied. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Day 84
Population: Safety analysis set with available data at both time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale | 2.8 (1.84) | 2.3 (3.51) | 3.2 (1.56) | 1.8 (1.71) | 2.3 (1.95) | 2.3 (1.50) | 2.4 (1.38) | 2.0 (1.41)

9. Secondary Outcome: Change From Baseline in Submental Skin Laxity Grades (SMSLG)
Description: Skin laxity assessment was based on clinical evaluation and palpation of the submental area on the following scale: 1 = no laxity; 2 = mild laxity; 3 = moderate laxity; 4 = severe laxity. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Day 84
Population: Safety analysis set with available data at both time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
units on a scale | 0.2 (0.66) | 0.0 (0.00) | 0.1 (0.77) | 0.5 (0.58) | 0.3 (0.45) | 0.5 (0.58) | 0.3 (0.67) | 0.3 (0.50)

10. Secondary Outcome: Change From Baseline in Submental Fat Thickness
Description: Submental thickness was measured using caliper devices.
Time Frame: Baseline and Day 84
Population: Safety analysis set with available data at both time points
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
mm | -1.4 (1.67) | -2.3 (2.08) | -1.6 (2.34) | -0.3 (2.75) | -0.9 (3.77) | -2.3 (2.22) | -1.5 (3.33) | -2.8 (2.22)

11. Secondary Outcome: Patient Experience Questions
Description: Participants were asked to complete 3 patient experience questions, each answered as Yes or No:
  Given your experience in this study:
  1. Would you recommend this procedure to a friend?
  2. Would you agree to receive additional treatments?
  3. Has the treatment you received in this study affected your normal activities?
  The percentage of participants answering Yes on each question is reported.
Time Frame: Day 84
Population: Safety analysis set with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Number analyzed (Participants) | 16 | 3 | 16 | 4 | 16 | 4 | 18 | 4
percentage of participants
  Recommend to a Friend | 81 | 33 | 81 | 50 | 94 | 100 | 72 | 75
  Receive Additional Treatments | 81 | 67 | 88 | 50 | 94 | 100 | 78 | 100
  Normal Activity Affected | 13 | 0 | 13 | 0 | 19 | 0 | 11 | 25

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Paradigm 1 / Deoxycholic Acid Injection | Paradigm 1 / Placebo | Paradigm 2 / Deoxycholic Acid Injection | Paradigm 2 / Placebo | Paradigm 3 / Deoxycholic Acid Injection | Paradigm 3 / Placebo | Paradigm 4 / Deoxycholic Acid Injection | Paradigm 4 / Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/3 | 0/17 | 0/4 | 0/16 | 0/4 | 0/18 | 0/4
Other Adverse Events (participants affected / at risk) | 17/17 | 3/3 | 17/17 | 4/4 | 16/16 | 4/4 | 18/18 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paradigm 1 / Deoxycholic Acid Injection (N=17) | Paradigm 1 / Placebo (N=3) | Paradigm 2 / Deoxycholic Acid Injection (N=17) | Paradigm 2 / Placebo (N=4) | Paradigm 3 / Deoxycholic Acid Injection (N=16) | Paradigm 3 / Placebo (N=4) | Paradigm 4 / Deoxycholic Acid Injection (N=18) | Paradigm 4 / Placebo (N=4)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site alopecia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site anaesthesia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 13 | 0 | 14 | 0 | 11 | 1 | 8 | 2
Injection site dysaesthesia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 17 | 1 | 15 | 3 | 16 | 4 | 17 | 4
Injection site induration (General disorders) | 17 | 0 | 16 | 1 | 16 | 1 | 18 | 3
Injection site nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site oedema (General disorders) | 17 | 2 | 17 | 4 | 16 | 4 | 18 | 4
Injection site pain (General disorders) | 17 | 2 | 17 | 1 | 16 | 2 | 18 | 2
Injection site pruritus (General disorders) | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Injection site rash (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 2 | 0 | 1 | 0 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Study Agreement requires that the investigator or institution obtain written consent from Kythera prior to presenting and/or publishing results of this study.